CLINICAL TRIAL: NCT02523248
Title: Randomized Control Study Between Uvulopalatopharyngoplasty and Tonsillectomy in Adult Sleep Apnea Patients
Brief Title: Comparison Between UPPP and Tonsillectomy in Adult OSA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of Covid 19 pandemic situation delay in recruiting patients
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Danielle Friberg, Associate Professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/755-31/2
Record Dates: First submitted 2015-08-06; First posted 2015-08-14 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Tonsillectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tonsillectomy (Active Comparator): Tonsillectomy with cold steel
  Interventions: Procedure: tonsillectomy
- Uvulopalatopharyngoplasty (Active Comparator): Tonsillectomy and uvulopalatoplasty; using cold steel and single sutures of the palate and tonsillar pillars including palatopharyngeal muscle
  Interventions: Procedure: Uvulopalatopharyngoplasty

INTERVENTIONS:
Procedure: tonsillectomy — Tonsillectomy with cold steel
  Arms: Tonsillectomy
Procedure: Uvulopalatopharyngoplasty — Tonsillectomy and uvulopalatoplasty with cold steel and single sutures of the palate and tonsillar pillars including palatopharyngeal muscle
  Other Names: UPPP
  Arms: Uvulopalatopharyngoplasty

SUMMARY:
The aim of this randomized control study is to evaluate the effect of tonsillectomy with or without uvulopalatoplasty in treating adults with moderate to severe sleep apnea.

DETAILED DESCRIPTION:
Patients are after baseline PSG 1 included and randomized to either UPPP or TE. They are stratified according to tonsil size, those with size 2 in one group and those with 3-4 in another. They all undergo surgery within two months and thereafter PSG 2 after 6 months and PSG after 4 years. At PSG they fill in questionnaires and measurements of blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* AHI more than 15
* Friedmans stage I and II
* Tonsil size 2, 3 and 4
* BMI below 34
* Failed use of CPAP and dental device

Exclusion Criteria:

* Severe cardiovascular or neurological disease
* Prefers strongly one surgical method
* ASA IV

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2021-11 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Polysomnography: group differences of changes in apnea-hypopnea index (AHI) | 6 months
  measurements with inlab polysomnography

SECONDARY OUTCOMES:
Questionnaire: group differences of changes in daytime sleepiness | 6 months
  A validated questionnaire: Epworth sleepiness scale
Questionnaire: group differences in changes of general health | 6 months
  A validated question of self-reported health
Group differences in changes of blood pressure | 6 months
  Measurements of blood pressure the morning after inlab polysomnography

OTHER OUTCOMES:
Polysomnography: group differences of changes in apnea-hypopnea index (AHI) | 4 years
  measurements with inlab polysomnography
Questionnaire: group differences of changes in daytime sleepiness | 4 years
  A validated questionnaire: Epworth sleepiness scale
Questionnaire: group differences in changes of general health | 4 years
  A validated question of self-reported health
Questionnaire of pharyngeal side-effects pre-and postoperatively | 6 months
  Questionnaire with 10 questions of pharyngeal disturbances administrated before and 6 months after surgery
Postoperative bleeding complications | 6 months
  Patient charts how many days patients stayed at hospitals postoperatively, reoperations and medications

CONTACTS AND LOCATIONS:
Overall Officials: Bo Tideholm, MD, PhD, Study Director — Karolinska University Hospital, ORL dep
Locations (1):
- Orl dep, Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Derived] Sundman J, Nerfeldt P, Fehrm J, Bring J, Browaldh N, Friberg D. Effectiveness of Tonsillectomy vs Modified Uvulopalatopharyngoplasty in Patients With Tonsillar Hypertrophy and Obstructive Sleep Apnea: The TEAMUP Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2022 Dec 1;148(12):1173-1181. doi: 10.1001/jamaoto.2022.3432. PMID 36326742